CLINICAL TRIAL: NCT04418648
Title: A Phase II, Randomised Study of Toripalimab as Consolidation Therapy in Patients With Limited-Stage Small Cell Lung Cancer Who Have Not Progressed Following Concurrent Chemoradiotherapy
Brief Title: Study of Toripalimab for Limited-Stage Small Cell Lung Cancer Following Concurrent Chemoradiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Since the interim results of the ADRIATIC trial presented at the ASCO Annual Meeting in June 2024, the design of the control group is no longer consistent with current clinical practice.
Sponsor: Sun Yat-sen University (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Guangzhou Panyu Central Hospital (Other)
Responsible Party: Principal Investigator, Hui Liu, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-FXY-243
Record Dates: First submitted 2020-05-25; First posted 2020-06-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer Limited Stage
Keywords: Consolidation therapy; Toripalimab; Concurrent chemoradiotherapy
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toripalimab Consolidation (Experimental): Patients in experimental group will receive toripalimab consolidation (240 mg) via iv infusion Q3W.
  Interventions: Drug: Toripalimab
- Observation (No Intervention): Patients in this group will receive observation.

INTERVENTIONS:
Drug: Toripalimab — Toripalimab consolidation (240 mg) via iv infusion once every 3 weeks. Administration of toripalimab will commence on Day 1 following randomisation to toripalimab after confirmation of eligibility and will continue on a Q3W schedule for a maximum duration of 6 months.
  Arms: Toripalimab Consolidation

SUMMARY:
The phase II, randomised study is to explore the efficacy and safety of toripalimab as consolidation therapy in patients with limited-stage small cell lung cancer who have not progressed following concurrent chemoradiation therapy

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures;
* Male or female aged 18-75 years;
* Histologically- or cytologically-documented SCLC;
* Stage I-III (AJCC/UICC 8th TNM Staging), with all lesions can be included in a tolerable radiotherapy field (limited-stage);
* Previous thoracic radiotherapy (45 Gy twice daily or 60-66 Gy once daily) and concurrent etoposide and platinum for four cycles; Dose coverage ≥ 85% of PTV-GTV. Radiotherapy started before the completion of the third cycle of chemotherapy;
* CR, PR or SD after concurrent chemoradiotherapy (RECIST v1.1);
* PCI is allowed and should be completed within 90 days after the completion of chemoradiotherapy;
* Randommization shoud be completed within 90 days after the completion of chemoradiotherapy;
* Life expectancy ≥12 weeks;
* World Health Organization (WHO) Performance Status of 0 or 1;
* Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients within 7 days before the use of study drug (HCG has a minimum sensitivity of 25 IU/L or equivalent);
* Women must be non-breastfeeding;
* Women of reproductive age (WOCBP) must agree to comply with the contraceptive method during the study toripalimab treatment and for a period of 3 months following the last administration of the study treatment (i.e., 30 days [ovulation cycle] plus approximately 5 half-lives of the study drug);
* Men who have sex with WOCBP must agree to comply with the contraceptive method during the study nivolumab treatment and for 5 months after the last administration of the study treatment (i.e. 90 days [sperm renewal cycle] plus approximately 5 half-lives of the study drug);
* Spermless men do not have to comply with contraceptive requirements. WOCBP who continues to be asexual with the opposite sex does not have to comply with contraceptive requirements, but must still undergo the pregnancy tests described in this section;
* Adequate organ and marrow function as defined below:

  1. Forced expiratory volume in 1 second (FEV1) ≥ 800ml;
  2. Absolute neutrophil count ≥1.5 x 10^9/L (1500 per mm3);
  3. Platelets ≥100 x 10^9/L (100,000 per mm3);
  4. Haemoglobin ≥ 9.0 g/dL (5.59 mmol/L);
  5. Serum creatinine clearance (CL) ≥ 50 mL/min by the Cockcroft-Gault formula (Cockcroft and -Gault 1976);
  6. Serum bilirubin ≤1.5 x upper limit of normal (ULN);
  7. Aspartate Transaminase (AST) and Alanine Transaminase (ALT) ≤ 2.5 x ULN.

Exclusion Criteria:

* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study;
* Mixed small cell and non-small cell lung cancer histology;
* Extensive-stage SCLC;
* Histologically-confirmed malignant pleural or pericardial effusion;
* Sequential chemoradiotherapy, or radiotherapy did not start before the completion of the third cycle of chemotherapy;
* Progressive disease after concurrent chemoradiotherapy (RECIST v1.1) and before randomization;
* Prior use of surgery, radiotherapy or chemotherapy for SCLC, with the exceptions of thoracic concurrent chemoradiotherapy and PCI;
* Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy will be excluded from randomization;
* Patients with Grade ≥2 pneumonitis from prior chemoradiation therapy will be excluded from randomization;
* Current or prior use of immunosuppressive medication within 28 days before the first dose of toripalimab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the previous chemoradiotherapy for SCLC is allowed;
* Prior exposure to any anti-programmed cell death protein(PD)-1 or anti-PD-L1 antibody;
* Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access);
* Active or prior documented autoimmune disease within the past 2 years including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granuloma, Sjogren's syndrome, Guillain Barre syndrome or multiple sclerosis;
* History of primary immunodeficiency;
* History of organ transplant that requires therapeutic immunosuppression;
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Bazett's Correction;
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, hepatitis C , human immunodeficiency virus (HIV), or patients with positive HBsAg and HBV-DNA > 500 IU/ml, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent;
* Known history of tuberculosis;
* Receipt of live attenuated vaccination within 30 days prior to study entry;
* History of another primary malignancy within 5 years prior to study entry, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ, breast intraductal carcinoma in situ or localized prostate cancer;
* Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control;
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the toripalimab or interpretation of patient safety or study results;
* Any condition that, in the opinion of the investigator, not suitable for study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | 2 years
  Time from the date of randomisation until death from any cause or first documented disease progression determined by RECISIT v1.1

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Time from the date of randomisation until death from any cause
Objective Response Rate | 2 years
  Best overall response (CR or PR) rate determined by RECISIT v1.1 across all assessment time-points during the period from randomisation to termination of protocol specific treatment
Duration of Response | 2 years
  Time from the date of first documented response of CR or PR until first documented progression or death, determined by RECISIT v1.1
Adverse Event | 2 years
  Number of participants with treatment-related adverse events determined by CTCAE v4.0
Quality of Life (EORTC QLQ-C30) | 2 years
  Quality of life score assessed by Quality of Life Questionnaire-Core 30 proposed by The European O-rganization for Reasearch and Treatment of Cancer. EORTC QLQ-C30 contained 30 items. Items 29 and 30 are rated on a scale of 1 to 7. The other items are divided into four grades: totally not, a little bit, a lot and very much, and scored on a scale of 1 to 4. For functional and overall health domain, a higher score refers to a better life quality; for symptom domain, a higher score refers to a worse life quality.
Quality of Life (EORTC QLQ-LC13) | 2 years
  Quality of life score assessed by Quality of Life Questionnare-Lung Cancer 13 proposed by The European O-rganization for Reasearch and Treatment of Cancer. EORTC QLQ-LC13 contained 13 items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. Each item is scored on a scale 0 to 100, where 0 indicates no symptoms and 100 indicates the worst possible symptoms.
ECOG performance status | 2 years
  Performance status score assessed by Zubrod-ECOG-WHO method, range 0-5. A higher score refers to a worse quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China